CLINICAL TRIAL: NCT02507024
Title: The ANCA Vasculitis Questionnaire (AAV-PRO©)
Acronym: AAV-PRO
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Collaborators: University of Oxford (Other); University of South Florida (Other)
Responsible Party: Sponsor
Other Study IDs: VCRC 5537
Record Dates: First submitted 2015-07-15; First posted 2015-07-23 (Estimated); Last update posted 2017-05-04 (Actual); Status verified 2017-05

CONDITIONS: Eosinophilic Granulomatosis With Polyangiitis (Churg-Strauss) (EGPA); Churg-Strauss Syndrome (CSS); Granulomatosis With Polyangiitis (Wegener's) (GPA); Wegener Granulomatosis (WG); Microscopic Polyangiitis (MPA); ANCA-Associated Vasculitis (AAV); Vasculitis
MeSH Terms: conditions — Churg-Strauss Syndrome; Granulomatosis with Polyangiitis; Microscopic Polyangiitis; Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis; Vasculitis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Intervention: The online questionnaire includes questions about how ANCA-associated vasculitis effects patients quality of life.
  Interventions: Other: Online questionnaire

INTERVENTIONS:
Other: Online questionnaire

SUMMARY:
The aim of this project is to develop a disease specific patient reported outcome measure (PROM) for patients with AAV (the AAV-PRO). Investigators are developing and validating a questionnaire to assess quality of life in patients with ANCA-associated vasculitis (AAV). Patients with AAV have inflammation in the small blood vessels leading to involvement of a range of organs and can suffer from ongoing disease activity or treatment side effects. Quality of life can be measured by patient reported outcome measures (PROMs).

DETAILED DESCRIPTION:
Patients with ANCA-associated vasculitis have inflammation in the small vessels that impact a range of organs and Investigators understand that patients may suffer ongoing disease activity, as well as side effects from the treatments. Assessing patients quality of life can be an important tool for conducting clinical trials for new treatments and medications.

Quality of life can be measured by questionnaires called "patient reported outcome measures" (PROM). What is a patient-reported outcome? Patient-reported outcomes, or PROs, are patients' feedback on what they are feeling or what they are able to do as participants are dealing with a chronic disease . Patient-reported outcomes are important because they provide doctors and researchers information about patients' quality of life. Questionnaires can be designed to measure specific PROs that are of specific importance to a disease and can provide much needed information on evaluating the effectiveness of health care. The aim of this survey is to develop a disease specific patient reported outcome measure, or PROM, for patients with AAV.

A small group of Investigators and Patient-Partners developed this survey for people with ANCA-associated vasculitis (the AAV-PRO). Investigators will invite patients with AAV to complete the questionnaire they have designed, called the AAV-PRO. By analysing how people fill in the questionnaire, Investigators will be able to find out how well the questions work, and whether they need to ask all of them.

ELIGIBILITY:
Inclusion Criteria:

* Registered in the Vasculitis Patient-Powered Research Network (V-PPRN)
* Patients greater than 18 years of age
* Diagnosis of ANCA-associated vasculitis including: Eosinophilic Granulomatosis with Polyangiitis (also called Churg-Strauss Syndrome), Granulomatosis with Polyangiitis (also called Wegener's granulomatosis or GPA), Microscopic Polyangiitis (MPA)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with AAV participating in the V-PPRN.
Sampling Method: Non-Probability Sample
Enrollment: 280 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Completion of AAV-PRO questionnaire. | 6 months
  Analysis of how people fill in the questionnaire to determine if these specific questions work, and whether we need to ask all of them.

CONTACTS AND LOCATIONS:
Overall Officials: Joanna Robson, MD, Principal Investigator — University of Oxford; Peter A Merkel, MD, MPH, Study Director — University of Pennsylvania
Locations (2):
- United States (2):
  - University of South Florida, Tampa, Florida
  - University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: V-PPRN Study Overview — http://www.vpprn.org/AAV-PRO